CLINICAL TRIAL: NCT05522179
Title: Nutritional Supplements to Support Recovery After Foot Surgery - A Pilot Study
Brief Title: Nutritional Supplements and Foot Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: NutraHeal (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: NH001
Record Dates: First submitted 2022-08-18; First posted 2022-08-30 (Actual); Last update posted 2023-08-01 (Actual); Status verified 2023-07

CONDITIONS: Foot Injuries and Disorders
Keywords: Nutritional supplements
MeSH Terms: conditions — Foot Injuries; Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- NutraHeal (Experimental): NutraHeal™ is a nutritional supplement that contains 7.5 micrograms (300 IU) of Vitamin D3, 80 mg of Calcium as Calcium Hydroxymethylbutyrate Monohydrate, 7.5 mg of Zinc, 600 mg of Calcium Hydroxymethylbutyrate Monohydrate, and 45 mg of Bromelain.
  Interventions: Dietary Supplement: NutraHeal
- NutraHeal Plus (Experimental): NutraHeal Plus™ is a nutritional supplement that contains 80 mg of Calcium as Calcium Hydroxymethylbutyrate Monohydrate, 7.5 mg of Zinc, 600 mg of Calcium Hydroxymethylbutyrate Monohydrate, 45 mg of Bromelain, and 7.5 mg of reduced Nicotinamide Adenine Dinucleotide (NADH).
  Interventions: Dietary Supplement: NutraHeal Plus
- Standard of Care (No Intervention): Receive standard of care for 1 week prior to surgery and 3 weeks after foot surgery.

INTERVENTIONS:
Dietary Supplement: NutraHeal — Receive NutraHeal (2 capsules twice a day) as a dietary supplement beginning 1 week prior to surgery and extending to 3 weeks after foot surgery.
  Arms: NutraHeal
Dietary Supplement: NutraHeal Plus — Receive NutraHeal Plus (2 capsules twice a day) as a dietary supplement beginning 1 week prior to surgery and extending to 3 weeks after foot surgery.
  Arms: NutraHeal Plus

SUMMARY:
This is a prospective randomized trial wherein participants will be assigned to NutraHeal™, NutraHeal Plus™, or standard of care for 1 week prior to foot surgery and 3 weeks after surgery. The central hypothesis is that among patients undergoing surgery, nutritional supplements that maintain energy production, muscle structure, immune function, and response to pain will support recovery from surgery.

DETAILED DESCRIPTION:
Over a 6 month period the investigators will enroll 45 male and female patients undergoing foot surgery. This is a prospective randomized trial and participants will be assigned to NutraHeal™ (n=15), NutraHeal Plus™ (n=15), or standard of care (n=15) for 1 week prior to surgery and 3 weeks after surgery. NutraHeal™ is a nutritional supplement that contains 7.5 micrograms (300 IU) of Vitamin D3, 80 mg of Calcium as Calcium Hydroxymethylbutyrate Monohydrate, 7.5 mg of Zinc, 600 mg of Calcium Hydroxymethylbutyrate Monohydrate, and 45 mg of Bromelain. NutraHeal Plus™ is a nutritional supplement that contains 80 mg of Calcium as Calcium Hydroxymethylbutyrate Monohydrate, 7.5 mg of Zinc, 600 mg of Calcium Hydroxymethylbutyrate Monohydrate, 45 mg of Bromelain, and 7.5 mg of reduced Nicotinamide Adenine Dinucleotide (NADH). Patients randomized to standard of care will not receive any of the ingredients in NutraHeal™ or NutraHeal Plus™.

The foot surgeon will evaluate the patient for wound healing time, healing quality, erythema and new tissue quality, using a Likert rating scale against expected results from -4 (much worse) to +4 (much better) including the expected reference grade of zero (0). Wound healing will be assessed at 1 and 3 weeks after surgery. Patients will document medication compliance (day of surgery, 1 and 3 weeks after surgery), pain medication use (baseline, on the day of surgery and at 1 and 3 weeks after surgery) and rate overall satisfaction (5-point scale (1 = excellent; 2 = good; 3 = moderate; 4 = sufficient; 5 = unsatisfactory) at 3 weeks after surgery). Patients will also complete the PROMIS-29 instrument at baseline, the day of surgery, and at 1 and 3 weeks after surgery).

ELIGIBILITY:
Inclusion Criteria:

* ≥ 20 years of age
* Undergoing foot surgery (matrixectomy (ingrown toenail removal) and wart removal)

Exclusion Criteria:

* > 80 years of age
* Pregnant patients or those anticipating pregnancy in the 1 month study period
* Allergic to pineapple
* Treated with oral anticoagulation
* Currently receiving Bromelain, Hydroxymethylbutyrate Monohydrate (HMB), reduced Nicotinamide Adenine Dinucleotide (NADH), Vitamin D3, or Zinc.
* Alcoholism (>2 drinks/day)
* Insulin Dependent Diabetes
* Hepatic insufficiency (prior known liver function tests > 1.5 times the upper limit of normal)
* Renal failure (prior known creatinine > 2.0 mg/dl)
* Severe pulmonary disease (requiring home oxygen therapy)
* Psychiatric illness requiring therapy (DSM-V thought disorders, recurrent major depressive disorder)

Ages: 20 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 46 (Actual)
Dates: Start 2022-08-29 (Actual); Primary Completion 2023-03-17 (Actual); Study Completion 2023-07-30 (Actual)

PRIMARY OUTCOMES:
Wound Healing at 3 weeks after surgery | 3 weeks after surgery.
  Wound healing (time, healing quality, erythema and new tissue quality), using a Likert rating scale against expected results from -4 (much worse) to +4 (much better) including the expected reference grade of zero (0). Positive scores are a better outcome.

SECONDARY OUTCOMES:
Pain Intensity | Baseline, the day of surgery, and at 1 and 3 weeks after surgery.
  Average pain intensity over previous 7 days as recorded in PROMIS-29. Pain intensity is graded on a visual analog scale from 0 (no pain) to 10 (worst imaginable pain). Higher scores mean a worse outcome.
Pain Interference | Baseline, the day of surgery, and at 1 and 3 weeks after surgery.
  Average pain interference over previous 7 days as recorded in PROMIS-29. Pain interference is graded on a scale of 1-5 (1 = Not at all, 2 = A little bit, 3 = Somewhat, 4 = Quite a bit, 5 = Very much). Higher scores mean a worse outcome.
Fatigue | Baseline, the day of surgery, and at 1 and 3 weeks after surgery.
  Fatigue over previous 7 days as recorded in PROMIS-29. Fatigue is graded on a scale of 1-5 (1 = Not at all, 2 = A little bit, 3 = Somewhat, 4 = Quite a bit, 5 = Very much). Higher scores mean a worse outcome.
Wound Healing at 1 week after surgery | 1 week after surgery
  Wound healing (time, healing quality, erythema and new tissue quality), using a Likert rating scale against expected results from -4 (much worse) to +4 (much better) including the expected reference grade of zero (0). Positive scores are a better outcome.

OTHER OUTCOMES:
Sleep Disturbance | Baseline, the day of surgery, and at 1 and 3 weeks after surgery.
  Sleep disturbance over previous 7 days as recorded in PROMIS-29. Sleep quality is assessed on a scale of 1-5 (1 = very good, 2 = good, 3= fair, 4 = poor, 5 = very poor). Higher scores indicate a worse outcome.
Physical Function | Baseline, the day of surgery, and at 1 and 3 weeks after surgery.
  Physical function as recorded in PROMIS-29. Physical function is assessed on a scale of 1-5 (1 = without any difficulty, 2 = with a little difficulty, 3= with some difficulty, 4 = with much difficulty, 5 = unable to do). Higher scores indicate a worse outcome.
Patient Satisfaction | 3 weeks after surgery.
  Overall satisfaction with 1) use of the nutritional supplements and 2) wound healing. Satisfaction is assessed on a scale of 1-5 (1 = excellent, 2 = good, 3 = moderate, 4 = sufficient, 5 = unsatisfactory). Higher scores indicate a worse outcome.

CONTACTS AND LOCATIONS:
Overall Officials: Lenore Moyer, DPM, Principal Investigator — Advanced Regional Center for Ankle and Foot Care
Locations (3):
- United States (3):
  - Advanced Regional Center for Ankle and Foot Care, Altoona, Pennsylvania
  - Advanced Regional Center for Ankle & Foot Care, Ebensburg, Pennsylvania
  - Advanced Regional Center for Ankle & Foot Care, State College, Pennsylvania

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Wischmeyer PE, Carli F, Evans DC, Guilbert S, Kozar R, Pryor A, Thiele RH, Everett S, Grocott M, Gan TJ, Shaw AD, Thacker JKM, Miller TE, Hedrick TL, McEvoy MD, Mythen MG, Bergamaschi R, Gupta R, Holubar SD, Senagore AJ, Abola RE, Bennett-Guerrero E, Kent ML, Feldman LS, Fiore JF Jr; Perioperative Quality Initiative (POQI) 2 Workgroup. American Society for Enhanced Recovery and Perioperative Quality Initiative Joint Consensus Statement on Nutrition Screening and Therapy Within a Surgical Enhanced Recovery Pathway. Anesth Analg. 2018 Jun;126(6):1883-1895. doi: 10.1213/ANE.0000000000002743. PMID 29369092
- [Background] Gillis C, Wischmeyer PE. Pre-operative nutrition and the elective surgical patient: why, how and what? Anaesthesia. 2019 Jan;74 Suppl 1:27-35. doi: 10.1111/anae.14506. PMID 30604414
- [Background] Paddon-Jones D, Campbell WW, Jacques PF, Kritchevsky SB, Moore LL, Rodriguez NR, van Loon LJ. Protein and healthy aging. Am J Clin Nutr. 2015 Jun;101(6):1339S-1345S. doi: 10.3945/ajcn.114.084061. Epub 2015 Apr 29. PMID 25926511
- [Background] MacKay D, Miller AL. Nutritional support for wound healing. Altern Med Rev. 2003 Nov;8(4):359-77. PMID 14653765
- [Background] Brien S, Lewith G, Walker A, Hicks SM, Middleton D. Bromelain as a Treatment for Osteoarthritis: a Review of Clinical Studies. Evid Based Complement Alternat Med. 2004 Dec;1(3):251-257. doi: 10.1093/ecam/neh035. Epub 2004 Oct 6. PMID 15841258
- [Background] Howat RC, Lewis GD. The effect of bromelain therapy on episiotomy wounds--a double blind controlled clinical trial. J Obstet Gynaecol Br Commonw. 1972 Oct;79(10):951-3. doi: 10.1111/j.1471-0528.1972.tb12194.x. No abstract available. PMID 4563795
- [Background] Landi F, Calvani R, Picca A, Marzetti E. Beta-hydroxy-beta-methylbutyrate and sarcopenia: from biological plausibility to clinical evidence. Curr Opin Clin Nutr Metab Care. 2019 Jan;22(1):37-43. doi: 10.1097/MCO.0000000000000524. PMID 30489401
- [Background] Ekinci O, Yanik S, Terzioglu Bebitoglu B, Yilmaz Akyuz E, Dokuyucu A, Erdem S. Effect of Calcium beta-Hydroxy-beta-Methylbutyrate (CaHMB), Vitamin D, and Protein Supplementation on Postoperative Immobilization in Malnourished Older Adult Patients With Hip Fracture: A Randomized Controlled Study. Nutr Clin Pract. 2016 Dec;31(6):829-835. doi: 10.1177/0884533616629628. Epub 2016 Jul 9. PMID 26965178
- [Background] Lautrup S, Sinclair DA, Mattson MP, Fang EF. NAD+ in Brain Aging and Neurodegenerative Disorders. Cell Metab. 2019 Oct 1;30(4):630-655. doi: 10.1016/j.cmet.2019.09.001. PMID 31577933
- [Background] Yoshino M, Yoshino J, Kayser BD, Patti GJ, Franczyk MP, Mills KF, Sindelar M, Pietka T, Patterson BW, Imai SI, Klein S. Nicotinamide mononucleotide increases muscle insulin sensitivity in prediabetic women. Science. 2021 Jun 11;372(6547):1224-1229. doi: 10.1126/science.abe9985. Epub 2021 Apr 22. PMID 33888596
- [Background] Iglar PJ, Hogan KJ. Vitamin D status and surgical outcomes: a systematic review. Patient Saf Surg. 2015 Apr 30;9:14. doi: 10.1186/s13037-015-0060-y. eCollection 2015. PMID 25926889
- [Background] Krasowska K, Skrobot W, Liedtke E, Sawicki P, Flis DJ, Dzik KP, Libionka W, Kloc W, Kaczor JJ. The Preoperative Supplementation With Vitamin D Attenuated Pain Intensity and Reduced the Level of Pro-inflammatory Markers in Patients After Posterior Lumbar Interbody Fusion. Front Pharmacol. 2019 May 22;10:527. doi: 10.3389/fphar.2019.00527. eCollection 2019. PMID 31191300
- [Background] Bonaventura P, Benedetti G, Albarede F, Miossec P. Zinc and its role in immunity and inflammation. Autoimmun Rev. 2015 Apr;14(4):277-85. doi: 10.1016/j.autrev.2014.11.008. Epub 2014 Nov 24. PMID 25462582
- [Background] Lin PH, Sermersheim M, Li H, Lee PHU, Steinberg SM, Ma J. Zinc in Wound Healing Modulation. Nutrients. 2017 Dec 24;10(1):16. doi: 10.3390/nu10010016. PMID 29295546